CLINICAL TRIAL: NCT03965195
Title: Comparative Effectiveness of Recombinant Versus Standard Dose Quadrivalent Influenza Vaccine in U.S. Nursing Homes
Brief Title: Recombinant Influenza Vaccination in U.S. Nursing Homes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Brown University (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INSI-201902
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Influenza; Influenza -Like Illness; Influenza, Human
Keywords: Influenza; Vaccine; Vaccination; Nursing Home; Respiratory-Related Hospitalizations; Cluster Randomized Trial; MACE (Major Adverse Cardiovascular Event); Cardiorespiratory-Related Hospitalizations; All-Cause Hospitalization
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RIV4 (Experimental): Nursing homes randomized to receive quadrivalent recombinant influenza vaccine (Flublok) for the residents and staff
  Interventions: Biological: Recombinant Influenza Vaccine
- IV4 (Active Comparator): Nursing homes randomized to receive standard dose quadrivalent influenza vaccine for the residents and staff
  Interventions: Biological: Standard Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Recombinant Influenza Vaccine — Nursing home residents and staff 18 years and older are allocated to receive quadrivalent recombinant influenza vaccine.
  Other Names: Flublok; RIV4
  Arms: RIV4
Biological: Standard Dose Quadrivalent Influenza Vaccine — Nursing home residents and staff 18 years and older are allocated to receive standard dose quadrivalent influenza vaccine
  Other Names: IV4
  Arms: IV4

SUMMARY:
Based on recent evidence on the mutation of the A/H3N2 strain in egg-grown vaccine, the investigators will study the quadrivalent recombinant influenza vaccine (RIV4, Flublok) compared to the standard dose quadrivalent vaccine (IV4) in a cohort of long-stay NH residents with a primary endpoint of all-cause hospitalization.

DETAILED DESCRIPTION:
A study sample goal of 1000 U.S. NHs, housing approximately 112,000 overall residents and 92,000 over the age of 65 years, of whom 64,500 are long-stay NH residents, will be recruited for each of the 2019-20 and 2020-21 influenza seasons. Participating facilities will be randomly allocated in a 1:1 ratio to RIV4 or IV4 vaccine for their residents. Also, all staff must be offered the same vaccine in both allocation groups, in order to eliminate differences in transmission of influenza through staff to residents related to differences in vaccine-related protection of staff and will reduce heterogeneity between clusters. The Minimum Data Set from the NH resident assessment instrument will be evaluated from all evaluable facilities meeting inclusion criteria and will be cross-referenced to Medicare claims and drug use data.

ELIGIBILITY:
Inclusion Criteria:

* Medicare-certified NHs with at least 50 long-stay residents ≥ 18 years of age
* Facilities with at least 80% of their long-stay population ≥ 65 years of age or at least 70 long stay residents ≥ 65 years of age that make up ≥ 45% of their total number of beds

Exclusion Criteria:

* Hospital-based facilities
* Facilities where Fluzone High-Dose or Fluad was used in the previous influenza season (2018-19 or 2019-20), or who's leadership plans to use one of these vaccines in the 2019- 2020 or 2020-21 season
* Facilities not submitting MDS data
* Facilities not in one of the 50 U.S. states

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1989 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Differences in all-cause hospitalization rates during the 2019-20 and 2020-21 influenza seasons | Up to 8 months each influenza season
  To determine the differences in all-cause hospitalization rates during the 2019-20 and 2020-21 influenza seasons experienced by all long-stay nursing home residents 18 years of age and older in facilities randomized to offer either quadrivalent recombinant influenza vaccine (RIV4) or standard dose quadrivalent influenza vaccine (IV4).

SECONDARY OUTCOMES:
Differences in each pneumonia and influenza-related hospitalization rates | Up to 8 months each influenza season
  To determine the differences in each pneumonia and influenza-related hospitalization rates during the 2019-20 and 2020-21 influenza seasons experienced by long-stay nursing home residents in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in pneumonia-related hospitalization rates | Up to 8 months each influenza season
  To determine the differences in each pneumonia-related hospitalization rates during the 2019-20 and 2020-21 influenza seasons experienced by long-stay nursing home residents in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in major adverse cardiovascular event-related (MACE) hospitalization rates | Up to 8 months each influenza season
  To determine the differences in each major adverse cardiovascular event-related (MACE) hospitalization rates during the 2019-20 and 2020-21 influenza seasons experienced by long-stay nursing home residents in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in cardiorespiratory-related hospitalization rates | Up to 8 months each influenza season
  To determine the differences in long-stay residents' cardiorespiratory-related hospitalization rates each season and across two seasons in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in ICU stay | Up to 8 months each influenza season
  To determine the differences in long-stay residents' ICU stay each season and across two seasons in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in mortality rates | Up to 8 months each influenza season
  To determine the differences in long-stay residents' mortality rates each influenza season and both seasons in facilities randomized to either RIV4 or IV4 for each, residents 18 years of age and older and those 65 years of age and older.
Differences in activities of daily living (ADL) function score | Up to 8 months each influenza season
  To determine the differences in long-stay residents' composite Activities of Daily Living (ADL) function score based on the MDS experienced during the influenza season by selected comorbidities and specific to respiratory illness, in facilities randomized to either RIV4 or IV4 combined over two seasons for each, residents 18 years of age and older and those 65 years of age and older.
Differences in facility-reported outbreaks | Up to 8 months each influenza season
  To determine differences in facility-reported outbreaks each season and across two seasons in facilities randomized to either RIV4 or IV4
Differences in all-cause hospitalization rates | Up to 8 months each influenza season
  To determine differences in long-stay residents' all-cause hospitalization rates as an interim exploratory analysis based on the Minimum Data Set 3.0 for each, residents 18 years of age and older and those 65 years of age and older.

CONTACTS AND LOCATIONS:
Overall Officials: H. Edward Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC; Stefan Gravenstein, MD, MPH, Principal Investigator — Insight Therapeutics, LLC
Locations (1):
- Insight Therapeutics, LLC, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McConeghy KW, Davidson HE, Canaday DH, Han L, Hayes K, Baier RR, Abul Y, Saade E, Mor V, Gravenstein S. Recombinant vs Egg-Based Quadrivalent Influenza Vaccination for Nursing Home Residents: A Cluster Randomized Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2452677. doi: 10.1001/jamanetworkopen.2024.52677. PMID 39745702